CLINICAL TRIAL: NCT04727879
Title: Beyond Analysis Of Blood Sample, to Approach Immunopathology of Polymyalgia Rheumatica on Shoulder Bursae's Biopsies: the BAOBAB Study
Brief Title: Immunopathology of Polymyalgia Rheumatica on Shoulder Bursae's Biopsies
Acronym: BAOBAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 29BRC20.0158
Record Dates: First submitted 2021-01-07; First posted 2021-01-27 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Polymyalgia Rheumatica
MeSH Terms: conditions — Polymyalgia Rheumatica | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PMR (Other): Patients with PMR will be offered biopsy of the synovial membrane with puncture of synovial fluid during cortisone infiltration for analgesic purposes. In case of associated peripheric arthritis, the patient will also be offered a joint fluid sample during a cortisonic infiltration for analgesic purposes, performed as part of routine care
  The study-specific examination that is not part of current practice is the synovial biopsy performed during the cortisonic infiltration procedure.
  Interventions: Procedure: Synovial membrane biopsy with puncture of synovial fluid; Procedure: Joint fluid sampling; Procedure: Blood sample
- Control (Other): Witnesses recruited into the orthopedic surgery department will be offered a synovial membrane biopsy during a shoulder surgery in the context of mechanical pathology.
  Interventions: Procedure: Synovial membrane biopsy with puncture of synovial fluid; Procedure: Blood sample

INTERVENTIONS:
Procedure: Synovial membrane biopsy with puncture of synovial fluid — The biopsy of the shoulder bursae will be carried out thanks to a device Tru-cut (Tru-Cut Biopsy Needle), minimally invasive, introduced, as during an infiltration, within the bursa serosa.
Procedure: Joint fluid sampling — In case of associated peripheric arthritis, the patient will also be offered a sample of joint fluid during a cortisonic infiltration for analgesic purposes, performed as part of routine care.
  Arms: PMR
Procedure: Blood sample — A blood sample taken during routine care and unused will also be collected from patients and controls for immunoassays.

SUMMARY:
The work carried out at the Brest University Hospital on serum immunological changes in patients with polymyalgia rheumatica (PMR) (based on clinical protocols TENOR, SEMAPHORE, THEN) made it possible to describe the changes in the distribution of lymphocyte subpopulations and cytokine levels during PPR, before and then under treatment compared to controls.

However, in systemic autoimmune or inflammatory pathologies, serum immunological mechanisms are rarely a reflection of intra-tissue mechanisms.

In the specific case of PMR, there are few data concerning muscular or joint immunological modifications. The investigators now wish to study the immunological modifications occurring at the tissue sites of interest, in particular in the shoulder bursae

ELIGIBILITY:
For everyone :

* Signed consent
* Patients over 50

Inclusion criteria :

For case patients:

* Addressed for PMR (diagnosis OR relapse)
* Score greater than or equal to 4 (without ultrasound criteria) or greater than or equal to 6 (with ultrasound criteria), according to the ACR / EULAR 2012 criteria for polymyalgia rheumatica, and suffering from bilateral scapular pain as well as an increased CRP level .
* Thickening of more than 2mm at least one shoulder bursae in ultrasound
* DAS-PPR> = 10

For witnesses:

- Shoulder surgery scheduled for mechanical pathology

Exclusion criteria :

For everyone :

* MRI with Gadolinium injection in the previous month- Clinical or paraclinical signs of giant cell arteritis
* Patient under protective measure or unable to consent
* Active cancer
* Active infection

For the cases:

- History of biotherapy treatment

For witnesses:

* History of inflammatory rheumatism
* Active inflammatory rheumatism

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-08-13 (Actual)

PRIMARY OUTCOMES:
IL-6 marking | Day 0
  The main evaluation criterion is the intensity of the tissue IL-6 marking on the subacromio-deltoid bursa sections using the Hyperion technique.

SECONDARY OUTCOMES:
Cytokinic (other than IL-6) infiltration of tissues | Day 0
Serum cytokine levels | Day 0
Cytokine levels in joint or synovial fluid | Day 0
Tissue distribution of lymphocyte subpopulations by using the Hyperion mass cytometer (analysis of the intensity of the markings) | Day 0
  Fragments of the synovial membrane taken from patients and controls will be sent to the pathology laboratory. They will be fixed and slides covering the inflammatory region of interest will be prepared. These slides will be marked with antibodies directed against: - CD20, CD27, CD38, CD24, CD21, CD95, CD23, IgM, Tbet for B lymphocytes; - CD3, CD4, CD8, CD25, CD45RA, CD62L, CD28, FoxP3, CCR7, CD45RO and Bcl-2 for T lymphocytes; - CD14, CD11b and CD11c for monocytes; - CD66b for granulocytes and coupled to heavy metals and analyzed by the Hyperion mass cytometer. The intensity of the markings will be analyzed using the usual Hyperion analysis techniques.
Serum distribution of lymphocyte subpopulations by using the HELIOS mass cytometer (analysis of the intensity of the markings) | Day 0
  Whole blood will be centrifuged and serum will be collected. Antibodies directed against: - CD20, CD27, CD38, CD24, CD21, CD95, CD23, IgM, Tbet for B lymphocytes; - CD3, CD4, CD8, CD25, CD45RA, CD62L, CD28, FoxP3, CCR7, CD45RO and Bcl-2 for T lymphocytes; - CD14, CD11b and CD11c for monocytes; - CD66b for granulocytes, aand Hnd coupled with heavy metals will be added to it before analysis by the HELIOS mass cytometer. The intensity of the markings will be analyzed using the usual HELIOS analysis techniques.
Analysis of immunosenescence markers in tissues by HYPERION technology | Day 0
  Analysis of membrane markers related to immunosenescence in percent of cells expressing the marker and in MFI (Mean fluorescence intensity) by hyperion technology.
Analysis of target molecules of treatments under study in PPR by ELISA technique | Day 0
  The target molecules of treatments under study in PPR (CTLA-4 for abatacept, janus kinases 1 and 2 for baricitinib) will be analyzed by ELISA techniques (concentration).
Analysis of target molecules of treatments under study in PPR by proteomic techniques | Day 0
  The target molecules of treatments under study in PPR (CTLA-4 for abatacept, janus kinases 1 and 2 for baricitinib) will be analyzed by protéomic techniques (cytometry, % of cells expressing the marker, MFI)
Complications of subacromio-deltoid purse in the 72h after biopsies : M1 phone call | Month 1
  The expected complications related to the synovial biopsy are:
  Pain at the biopsy site, Hematoma at the biopsy site, Functional impotence of the shoulder, on the biopsy side, greater than 72h, Hypoesthesia, dysesthesia at the biopsy site, Skin rash within 72h following the infiltration, Hypertensive surge documented within 72 hours of the infiltration, In case of pre-existing diabetes, diabetes imbalance within 72 hours of the infiltration.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Brest - Service de rhumatologie, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.